CLINICAL TRIAL: NCT01182376
Title: SOAR: Study Observing Antiarrhythmic Remodelling Using LGE-MRI
Acronym: SOAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Nassir F. Marrouche, MD, Associate Professor of cardiology, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB_00040931
Record Dates: First submitted 2010-08-11; First posted 2010-08-16 (Estimated); Results first posted 2016-02-19 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-01

CONDITIONS: Atrial Fibrillation
Keywords: Multaq; dronedarone; Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Dronedarone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Half of the patients will be assigned placebo.
  Interventions: Drug: Placebo
- Multaq® (dronedarone) (Experimental): Half of the patients will be prescribed dronedarone.
  Interventions: Drug: dronedarone

INTERVENTIONS:
Drug: dronedarone — Dronedarone will be prescribed by the patient's team according to established guidelines.
  Other Names: Multaq®
  Arms: Multaq® (dronedarone)
Drug: Placebo — Placebo will be administered by the patient's team according to established guidelines.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to demonstrate how dronedarone (Multaq®) may aid in the slowing of progression of left atrial and ventricular fibrosis in patients with atrial fibrillation as assessed by late gadolinium enhanced magnetic resonance imaging.

DETAILED DESCRIPTION:
BACKGROUND AND INTRODUCTION:

Atrial fibrillation (AF) arises as a result of a complex interaction between triggers, perpetuators and substrate. As early as 1995, Morillo et al have demonstrated that AF is associated with ultrastructural changes in myocytes. In animal models, alterations in myocytes after sustained AF resemble those of myocardial hybernation with a phenotypical adaptation towards a more fetal stage. Ultimately, these structural changes would lead to Calcium overload and metabolic stress, similar changes have been observed in humans. However, in humans, atrial dilatation and degenerative changes have been observed. Interstitial fibrosis (caused by deposits of collagen and fibronectin) is the prime cause of structural remodeling in left atrium (Boldt et al., 2004). It has been well established that fibrosis is a confounding clinical factor in causing AF (Kostin et al., 2002). But AF itself promotes fibrosis, which in turn leads to increased conduction heterogeneity within the atrial substrate resulting in further progression of AF (Everett,and Olgin, 2007).

The recent introduction of Late Gadolinium enhancement magnetic resonance imaging (LGE-MRI) sequence now allows for non-invasive assessment of the location and extent of arrhythmia related fibrosis.

Contrast enhancement occurs as a result of altered washout kinetics of gadolinium relative to normal surrounding tissue, which may reflect increased fibrosis or tissue remodeling of the myocardium. Our group has demonstrated the feasibility of a new LGE-MRI acquisition and processing protocol to detect fibrosis in the LA.

To date, no controlled trials evaluating the effect of antiarrhythmic drugs (AAD) and regression of left atrial fibrosis as assessed by LGE-MRI has been performed. We propose to use LGE-MRI to evaluate the effects of dronedarone vs. placebo on atrial and ventricular fibrosis. It has been shown that the success of catheter ablation procedure (which has been shown to be superior in terms of maintaining sinus rhythm in AF patients when compared to anti-arrhythmic drugs) is dependent upon the extent of fibrosis (Akoum et al., in prep). In AF patients with greater than 35% enhancement (percent left atrial fibrosis), the success of catheter ablation in reducing AF recurrence is greatly reduced. Hence for these patients, a drug that can control the progression of fibrosis and simultaneously provide respite from AF recurrence would be an extremely desirable prescription.

Multaq® is the chosen drug in this study because clinical trials (Hohnloser et al., 2009) have shown that it has the potential to reduce incidence of hospitalizations due to cardiovascular events by 25.5% and death in AF patients by 45%. We acknowledge the information that Dronedarone may be more prone to AF recurrence, however, it has a better safety profile with regards to thyroid and neurologic events and does not interfere with oral anticoagulants (Le Heuzey et al., 2010), which make dronedarone a more preferred antiarrhythmic drug to be used for this study. Furthermore, in patients who took dronedarone post cardioversion procedure to revert arrhythmia back to normal sinus rhythm (NSR), dronedarone has been shown to decrease AF recurrences (Le Heuzey et al., 2010).

OBJECTIVES:

Primary:

The primary objective of this study is to demonstrate how dronedarone may aid in the regression or slowing of progression of left atrial and ventricular fibrosis in patients with atrial fibrillation as assessed by LGE-MRI, using longitudinal data from a double-blinded, prospective study of patients diagnosed with atrial fibrillation over a twelve month follow up period.

Secondary:

* To study the effects of dronedarone in global parameters of myocardial remodeling such as right and left atrial volumes and right and left ventricular volumes.
* To study correlation between AF burden expressed as percentage of AF measured by an 8-day Holter Monitoring at three, six and twelve months post initiation.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 and older
* Must carry a diagnosis of Paroxysmal Atrial Fibrillation for 1 months or longer prior to being enrolled.
* AAD: Multaq® (dronedarone) candidate
* Patients have given informed consent

Exclusion Criteria:

* Patients who are unavailable to continue follow-up at the University of Utah outpatient clinic.
* Patients weighing >200 lbs (MR image efficacy decreases due to density)
* Prior RF Ablation treatment for atrial fibrillation
* Severe renal failure manifested by a chronic GFR of < 30 mL/min, or acute renal failure regardless of the GFR, until the renal function has stabilized. (Gadolinium contraindication)
* Enrollment in any other investigational trial for anti-arrhythmic therapy
* Any health related Gadolinium/MRI contraindications: Pacemaker devices, etc.
* Pregnant women
* Individuals with cognitive impairments who are unable to give informed consent
* Multaq® (dronedarone) contraindications:

  * NYHA Class IV heart failure or NYHA Class II - III heart failure with a recent decompensation requiring hospitalization or referral to a specialized heart failure clinic
  * Second- or third-degree atrioventricular (AV) block or sick sinus syndrome
  * Bradycardia < 50 bpm
  * Concomitant use of strong CYP 3A inhibitors, such as ketoconazole, itraconazole, voriconazole, cyclosporine, telithromycin, clarithromycin, nefazodone, and ritonavir
  * Concomitant use of drugs or herbal products that prolong the QT interval and might increase the risk of Torsade de Pointes, such as phenothiazine anti-psychotics, tricyclic antidepressants, certain oral macrolide antibiotics, and Class I and III antiarrhythmics
  * QTc Bazett interval ≥ 500 ms or PR interval > 280 ms
  * Severe hepatic impairment
  * Pregnant women
  * Nursing mothers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2010-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nassir F Marrouche, MD, Principal Investigator — University of Utah

REFERENCES:
- [Background] Swynghedauw B. Molecular mechanisms of myocardial remodeling. Physiol Rev. 1999 Jan;79(1):215-62. doi: 10.1152/physrev.1999.79.1.215. PMID 9922372
- [Background] Oral H, Pappone C, Chugh A, Good E, Bogun F, Pelosi F Jr, Bates ER, Lehmann MH, Vicedomini G, Augello G, Agricola E, Sala S, Santinelli V, Morady F. Circumferential pulmonary-vein ablation for chronic atrial fibrillation. N Engl J Med. 2006 Mar 2;354(9):934-41. doi: 10.1056/NEJMoa050955. PMID 16510747
- [Background] Lee SH, Tai CT, Hsieh MH, Tsai CF, Lin YK, Tsao HM, Yu WC, Huang JL, Ueng KC, Cheng JJ, Ding YA, Chen SA. Predictors of early and late recurrence of atrial fibrillation after catheter ablation of paroxysmal atrial fibrillation. J Interv Card Electrophysiol. 2004 Jun;10(3):221-6. doi: 10.1023/B:JICE.0000026915.02503.92. PMID 15133358
- [Background] Oral H, Knight BP, Ozaydin M, Tada H, Chugh A, Hassan S, Scharf C, Lai SW, Greenstein R, Pelosi F Jr, Strickberger SA, Morady F. Clinical significance of early recurrences of atrial fibrillation after pulmonary vein isolation. J Am Coll Cardiol. 2002 Jul 3;40(1):100-4. doi: 10.1016/s0735-1097(02)01939-3. PMID 12103262
- [Background] O'Donnell D, Furniss SS, Dunuwille A, Bourke JP. Delayed cure despite early recurrence after pulmonary vein isolation for atrial fibrillation. Am J Cardiol. 2003 Jan 1;91(1):83-5. doi: 10.1016/s0002-9149(02)03005-9. No abstract available. PMID 12505579
- [Background] Vasamreddy CR, Lickfett L, Jayam VK, Nasir K, Bradley DJ, Eldadah Z, Dickfeld T, Berger R, Calkins H. Predictors of recurrence following catheter ablation of atrial fibrillation using an irrigated-tip ablation catheter. J Cardiovasc Electrophysiol. 2004 Jun;15(6):692-7. doi: 10.1046/j.1540-8167.2004.03538.x. PMID 15175066
- [Background] Lo LW, Tai CT, Lin YJ, Chang SL, Wongcharoen W, Hsieh MH, Tuan TC, Udyavar AR, Hu YF, Chen YJ, Tsao HM, Chen SA. Mechanisms of recurrent atrial fibrillation: comparisons between segmental ostial versus circumferential pulmonary vein isolation. J Cardiovasc Electrophysiol. 2007 Aug;18(8):803-7. doi: 10.1111/j.1540-8167.2007.00848.x. Epub 2007 May 14. PMID 17504254
- [Background] Pappone C, Oreto G, Rosanio S, Vicedomini G, Tocchi M, Gugliotta F, Salvati A, Dicandia C, Calabro MP, Mazzone P, Ficarra E, Di Gioia C, Gulletta S, Nardi S, Santinelli V, Benussi S, Alfieri O. Atrial electroanatomic remodeling after circumferential radiofrequency pulmonary vein ablation: efficacy of an anatomic approach in a large cohort of patients with atrial fibrillation. Circulation. 2001 Nov 20;104(21):2539-44. doi: 10.1161/hc4601.098517. PMID 11714647
- [Background] Riley MJ, Marrouche NF. Ablation of atrial fibrillation. Curr Probl Cardiol. 2006 May;31(5):361-90. doi: 10.1016/j.cpcardiol.2006.01.002. PMID 16690376
- [Background] Wazni OM, Marrouche NF, Martin DO, Verma A, Bhargava M, Saliba W, Bash D, Schweikert R, Brachmann J, Gunther J, Gutleben K, Pisano E, Potenza D, Fanelli R, Raviele A, Themistoclakis S, Rossillo A, Bonso A, Natale A. Radiofrequency ablation vs antiarrhythmic drugs as first-line treatment of symptomatic atrial fibrillation: a randomized trial. JAMA. 2005 Jun 1;293(21):2634-40. doi: 10.1001/jama.293.21.2634. PMID 15928285
- [Background] Oakes RS, Badger TJ, Kholmovski EG, Akoum N, Burgon NS, Fish EN, Blauer JJ, Rao SN, DiBella EV, Segerson NM, Daccarett M, Windfelder J, McGann CJ, Parker D, MacLeod RS, Marrouche NF. Detection and quantification of left atrial structural remodeling with delayed-enhancement magnetic resonance imaging in patients with atrial fibrillation. Circulation. 2009 Apr 7;119(13):1758-67. doi: 10.1161/CIRCULATIONAHA.108.811877. Epub 2009 Mar 23. PMID 19307477
- [Background] Badger TJ, Oakes RS, Daccarett M, Burgon NS, Akoum N, Fish EN, Blauer JJ, Rao SN, Adjei-Poku Y, Kholmovski EG, Vijayakumar S, Di Bella EV, MacLeod RS, Marrouche NF. Temporal left atrial lesion formation after ablation of atrial fibrillation. Heart Rhythm. 2009 Feb;6(2):161-8. doi: 10.1016/j.hrthm.2008.10.042. Epub 2008 Nov 6. PMID 19187904
- [Background] Sinha AM, Schmidt M, Marschang H, Gutleben K, Ritscher G, Brachmann J, Marrouche NF. Role of left ventricular scar and Purkinje-like potentials during mapping and ablation of ventricular fibrillation in dilated cardiomyopathy. Pacing Clin Electrophysiol. 2009 Mar;32(3):286-90. doi: 10.1111/j.1540-8159.2008.02233.x. PMID 19272055
- [Background] Badger TJ, Adjei-Poku YA, Marrouche NF. MRI in cardiac electrophysiology: the emerging role of delayed-enhancement MRI in atrial fibrillation ablation. Future Cardiol. 2009 Jan;5(1):63-70. doi: 10.2217/14796678.5.1.63. PMID 19371204
- [Background] Weber KT, Weglicki WB, Simpson RU. Macro- and micronutrient dyshomeostasis in the adverse structural remodelling of myocardium. Cardiovasc Res. 2009 Feb 15;81(3):500-8. doi: 10.1093/cvr/cvn261. Epub 2008 Oct 3. PMID 18835843

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Half of the patients will be assigned placebo.
  dronedarone: Dronedarone will be prescribed by the patient's team according to established guidelines.
Period: Overall Study
Arm/Group | Placebo | Multaq® (Dronedarone)
Started | 15 | 18
Completed | 4 | 13
Not Completed | 11 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Multaq® (Dronedarone) | Total
Number analyzed (Participants) | 15 | 18 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 11 | 14
  >=65 years | 12 | 7 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 71 (8) | 64 (11) | 68 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 10 | 11 | 21
Pre-treatment left atrial fibrosis percentage [Mean (Standard Deviation); unit: percentage] — Percentage of left atrial fibrosis is determined using an MRI image of the acutal fibrotic tissue located on the surface of the left atrium. Proprietary software is used to calculate fibrosis percentage based on the image. Fibrosis percentage can range from 0% to 40%. As a rule, the higher the percentage the worse the cardiovascular outcome of the patient.
  percentage | 19.9 (.10) | 15.5 (.05) | 17.7 (.08)

OUTCOME MEASURES:

1. Primary Outcome: LA Fibrosis
Description: The change in left atrial fibrosis percentage, as measured on a scale, using MRI imaging, from baseline to the end of treatment.
Time Frame: baseline, 1 year
Population: The number of participants analyzed for both groups is less than the number enrolled due to patient attrition or poor MRI scans.
Measure: Mean (Standard Deviation); unit: percentage of fibrosis
Arm/Group | Placebo | Multaq® (Dronedarone)
Number analyzed (Participants) | 4 | 12
percentage of fibrosis | 24.6 (.07) | 16.8 (.05)

ADVERSE EVENTS:
Arm/Group | Placebo | Multaq® (Dronedarone)
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/18
Other Adverse Events (participants affected / at risk) | 11/15 | 6/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=15) | Multaq® (Dronedarone) (N=18)
Nausea (Gastrointestinal disorders) | 3 | 0
arrhythmias (Cardiac disorders) | 1 | 0 — Includes diagnosis of AF, long QT
non compliance (Social circumstances) | 5 | 2
other surgeries (Surgical and medical procedures) | 2 | 3 — Withdrawal due to other surgical procedures
drug interactions (General disorders) | 0 | 1 — concomittant drugs interacted with Multaq

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No